CLINICAL TRIAL: NCT01775202
Title: Cognitive Changes After Fast-track Colon Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lene Krenk (Other)
Responsible Party: Sponsor-Investigator, Lene Krenk, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-3-2012-FSP69
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Cogntive Changes After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This descriptive study aims to evalaute in a retrospective way the incidence of cogntive changes postoperatively after fast-track colon surgery at Hvidovre Hospital. This survey is based on chart reviews.

ELIGIBILITY:
Inclusion Criteria:

* > 59 years
* undergoing colon surgery at Hvidovre Hospital
* surgery and perioperative care in a fast-track setting

Exclusion Criteria:

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients > 60 years, undergoing fast-track colon surgery at Hvidovre Hospital during 2010-2012.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
cognitive change postoperatively based on chart review | during hospital stay (postoperative day 0-3)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of abdominal surgery (colon section) Hvidovre Hospital, Hvidovre, Denmark